CLINICAL TRIAL: NCT03518008
Title: Clinical Comparison of Two Daily Disposable Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLE383-C006
Record Dates: First submitted 2018-05-01; First posted 2018-05-08 (Actual); Results first posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Myopia; Refractive Errors
Keywords: soft contact lenses; vision; eyesight
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- DD T2, then Clariti 1 Day (Other): Verofilcon A contact lenses worn first, with somofilcon A contact lenses worn second. Each product worn bilaterally (in both eyes) for 1 week in a daily disposable modality.
  Interventions: Device: verofilcon A contact lenses; Device: somofilcon A contact lenses
- Clariti 1 Day, then DD T2 (Other): Somofilcon A contact lenses worn first, with verofilcon A contact lenses worn second. Each product worn bilaterally for 1 week in a daily disposable modality.
  Interventions: Device: verofilcon A contact lenses; Device: somofilcon A contact lenses

INTERVENTIONS:
Device: verofilcon A contact lenses — Investigational daily disposable soft contact lenses
  Other Names: DD T2
Device: somofilcon A contact lenses — Commercially available daily disposable soft contact lenses
  Other Names: clariti® 1 day; Clariti 1 Day

SUMMARY:
The purpose of this study is to evaluate the overall performance of investigational contact lenses (DD T2) when compared to clariti® 1 day contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Understand and sign an Informed Consent Form;
* Successful wear of daily disposable spherical soft contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months;
* Best-corrected visual acuity (BCVA) 20/25 or better in each eye;
* Willing to stop wearing habitual contact lenses for the duration of study participation;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Anterior segment infection, inflammation, or abnormality or disease that contraindicates contact lens wear, as determined by the Investigator;
* Use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the Investigator;
* Refractive, ocular, or intraocular surgery, as specified in the protocol;
* Eye condition or injury, as specified in the protocol;
* Current or history of intolerance, hypersensitivity, or allergy to any component of the study products;
* Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment;
* Use of topical ocular medications and artificial tear or rewetting drops requiring instillation during contact lens wear;
* Currently wearing clariti® 1 day contact lenses;
* Habitually wearing monovision or multifocal lenses during the last 3 months;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Research, Study Director — Alcon Research
Locations (1):
- Alcon Investigative Site, Maitland, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 investigative site located in the United States.
Pre-assignment Details: A total of 22 subjects signed informed consent to participate in the study. This reporting group includes all randomized and exposed subjects (22).
Groups:
- DDT2, Then Clariti 1 Day: Verofilcon A contact lenses worn first, with somofilcon A contact lenses worn second. Each product will be worn bilaterally (in both eyes) for 1 week in a daily disposable modality.
- Clariti 1 Day, Then DDT2: Somofilcon A contact lenses worn first, with verofilcon A contact lenses worn second. Each product will be worn bilaterally for 1 week in a daily disposable modality.
Period: Period 1, First Week of Wear
Arm/Group | DDT2, Then Clariti 1 Day | Clariti 1 Day, Then DDT2
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Period 2, Second Week of Wear
Arm/Group | DDT2, Then Clariti 1 Day | Clariti 1 Day, Then DDT2
Started | 11 | 11
Completed | 11 | 10
Not Completed | 0 | 1
Not completed — Family emergency | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study (Safety Analysis Set).
Groups:
- Overall: Verofilcon A and somofilcon A contact lenses worn during Period 1 and Period 2 in a crossover assignment, as randomized.
Arm/Group | Overall
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22
  Black or African American | 0
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Quality of Vision
Description: Overall quality of vision was measured as a subjective rating, collected binocularly on a scale of 1 (Poor) to 10 (Excellent). No inferences were made; therefore, no hypotheses were formulated.
Time Frame: Day 8, each product
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- DD T2: Verofilcon A contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2 for 1 week in a daily disposable modality
- Clariti 1 Day: Somofilcon A contact lenses worn bilaterally during Period 1 or Period 2 for 1 week in a daily disposable modality.
Arm/Group | DD T2 | Clariti 1 Day
Number analyzed (Participants) | 22 | 22
units on a scale | 9.2 (1.0) | 8.6 (1.5)

ADVERSE EVENTS:
Time Frame: Dispense through study completion, approximately 20 days
Description: An adverse event (AE) was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the investigational medical device. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol. Safety Analysis Set, based on treatment-specific exposure.
Groups:
- DD T2: All subjects exposed to verofilcon A contact lenses
- Clariti 1 Day: All subjects exposed to somofilcon A contact lenses
Arm/Group | DD T2 | Clariti 1 Day
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT03518008/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT03518008/SAP_001.pdf